CLINICAL TRIAL: NCT00229229
Title: Comparison of a Low Glycemic Load Diet With a Canada Food Guide Diet in the Management of Overweight Patients With Cardiovascular Disease
Brief Title: Comparison of 4 Diets in the Management of Overweight Patients With Vascular Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Queen's University (Other)
Responsible Party: Stephen LaHaye MD,FRCP, QUEEN'S UNIVERSITY
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DMED-793-04
Record Dates: First submitted 2005-09-09; First posted 2005-09-29 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Obesity; Cardiovascular Disease; Metabolic Syndrome
Keywords: Obesity; Cardiovascular Disease; Metabolic Syndrome; Canada Food Guide; Glycemic Index; Glycemic Load
MeSH Terms: conditions — Obesity; Cardiovascular Diseases; Metabolic Syndrome | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Other): Low glycemic load diet
  Interventions: Other: Low glycemic load diet
- 2 (Other): Canada Food Guide Diet
  Interventions: Other: Canada Food Guide Diet
- 3 (Other): Low glycemic index diet
  Interventions: Other: Low glycemic index diet
- 4 (Other): Low carbohydrate diet
  Interventions: Other: Low carbohydrate diet

INTERVENTIONS:
Other: Low glycemic load diet — A/A for 6 months intensive dietary intervention followed by a visit 1 year from enrolment
  Arms: 1
Other: Canada Food Guide Diet — A/A for 6 months intensive dietary intervention followed by a visit 1 year from enrolment
  Arms: 2
Other: Low glycemic index diet — A/A for 6 months intensive dietary intervention followed by a visit 1 year from enrolment
  Arms: 3
Other: Low carbohydrate diet — A/A for 6 months intensive dietary intervention followed by a visit 1 year from enrolment
  Arms: 4

SUMMARY:
Type 2 diabetes can be prevented by lifestyle changes in high-risk subjects. However, controversies exist on nutritional management of diabetes. Recent data suggests that glucose and insulin responses are affected by not only the quality, but the quantity of carbohydrate consumed. This is referred to as glycemic load.

To date, there have not been any prospective randomized studies which examine the utility of a low glycemic load diet.

The purpose of the proposed study is to compare the effectiveness of a Canada Food Guide Diet with a low glycemic load diet on blood sugar control in overweight type 2 diabetics.

DETAILED DESCRIPTION:
The primary objective of the proposed study is to compare the effectiveness of a low glycemic load diet with a Canada Food Guide Diet on weight loss in overweight subjects with cardiovascular disease.

The secondary objective of the proposed study is to compare the effectiveness of a low glycemic load diet with both a low glycemic index diet and a low carbohydrate diet on weight loss in overweight subjects with cardiovascular disease. The purpose of this portion of the study is to try to elucidate the relative contributions of the glycemic index and carbohydrate content to the overall effectiveness of a low glycemic load diet. Furthermore, through detailed analysis of actual dietary consumption, and correlation with subsequent weight loss, we hope to gain greater insight into the role of compliance on the success of the various dietary strategies. Restriction of caloric intake is necessary for weight loss regardless of the dietary strategy employed, however, long-term success depends ultimately on the ability of the patients to comply with the said diet. The success of a low glycemic load diet may lie in its superior effectiveness (greater compliance, less calorie consumption) rather than a greater efficacy per se.

A secondary analysis of the effects of all three diets (low glycemic load, low glycemic index and low carbohydrate) on modifying other metabolic factors will also be performed. In particular, the study will examine the effect of the three diets on lipid and fat metabolism, insulin resistance and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged 18 to 80 years
* BMI 25-40 kg/m2
* Documented Cardiovascular Disease as evidenced by one or more of the following:

  * Coronary atherosclerosis during coronary angiography
  * Documented myocardial infarction
  * Carotid atherosclerosis during carotid ultrasonography
  * Carotid atherosclerosis during CT angiography
  * Carotid atherosclerosis during MR angiography
  * Ischemic brain infarct documented on brain imaging studies

Exclusion Criteria:

* Documented Type I or II diabetes mellitus (as defined by the Canadian Diabetes Association 2003 Clinical Practice Guidelines for the Prevention and Management of Diabetes in Canada)
* Previous (<5 years ago) individual or group dietary counseling with a registered dietician
* Pregnant or lactating women
* Presence of clinically important hepatic or renal disease
* Inability to communicate effectively using the English language
* Enrollment in another study concurrently
* Inability to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2004-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To compare the effectiveness of a low glycemic load diet with a Canada Food Guide Diet on weight loss in overweight subjects with cardiovascular disease. | 1 year

SECONDARY OUTCOMES:
To compare the effectiveness of a low glycemic load diet with both a low glycemic index diet and a low carbohydrate diet on weight loss in overweight subjects with cardiovascular disease. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A LaHaye, MD, Principal Investigator — Vascular Disease Prevention and Research Centre
Locations (1):
- Vascular Disease Prevention and Research Centre, Kingston, Ontario, Canada